CLINICAL TRIAL: NCT02331524
Title: Exercise and Psychosocial-Based Interventions to Improve Daily Activity in Heart Failure
Brief Title: Interventions to Improve Daily Activity in Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grand Valley State University (Other)
Collaborators: Corewell Health West (Other)
Responsible Party: Principal Investigator, Michael J. Shoemaker, Associate Professor of Physical Therapy, Grand Valley State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-180-H
Record Dates: First submitted 2014-12-27; First posted 2015-01-06 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Heart Failure
Keywords: exercise; daily activity
MeSH Terms: conditions — Heart Failure; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control/Usual Care (No Intervention): Usual care only
- Activity Feedback and Encouragement (Experimental): Weekly Feedback about daily activity using the FitBit Zip
  Interventions: Behavioral: Activity Feedback and Encouragement
- Health Coaching/Home Exercise (Experimental): Weekly contact from physical therapist to develop and progress home exercise program and by health coach for goal setting and support
  Interventions: Other: Health Coaching/Home Exercise

INTERVENTIONS:
Behavioral: Activity Feedback and Encouragement — The Daily Activity Feedback/ Encouragement group will receive weekly feedback and encouragement regarding daily activity using the Fitbit Zip® for 3 months. Visual feedback and verbal encouragement will be provided. Visual feedback will provide graphics showing current and historical daily activity trends since the start of the intervention period. Subjects in the Feedback group will also receive standardized verbal feedback based upon the Fitbit Zip data. For example, subjects demonstrating a trend of increasing daily activity will be encouraged to "Continue what you are doing. You are doing great!"
  Arms: Activity Feedback and Encouragement
Other: Health Coaching/Home Exercise — The Health Coaching/Home Exercise group will receive 12 weekly health coaching and physical therapy visits for 3 months. Health coaching will be provided by a trained, highly experienced health and wellness coach. In-home health coaching sessions will be provided monthly (total of 3) with the remaining 9 sessions provided telephonically. Initial health coaching sessions will include the utilization of motivational interviewing to establish individualized, three-month goals related to symptoms, function, and/or daily activity, with subsequent sessions celebrating successes in and/or identifying barriers to achieving these goals.
  Arms: Health Coaching/Home Exercise

SUMMARY:
There are few studies that demonstrate how to best improve daily activity in people with heart failure (HF). Exercise alone has been shown to be ineffective, but other techniques such as daily activity feedback with encouragement or health coaching may be helpful. This research study will investigate two different treatment approaches for improving daily activity: 1) daily activity feedback and encouragement, and 2) health coaching with an individualized home exercise program. Both treatment approaches are hypothesized to result in improved daily activity compared to a control group.

DETAILED DESCRIPTION:
Few studies have been able to demonstrate intervention efficacy for improving daily activity in heart failure (HF). Exercise alone is ineffective, though psychosocial-based interventions including health coaching and daily activity feedback appear to be promising. Therefore, the primary purpose of the present proposed study is to investigate the effect of two different intervention approaches (1. daily activity feedback with associated encouragement, and 2. health coaching with an associated individualized home exercise program) on daily activity, exercise tolerance, HF-related health status, and lower extremity functional strength. A secondary purpose is to compare daily activity as recorded by Medtronic® implanted cardioverter defibrillator (ICDs) and cardiac resynchronization therapy (CRT) devices to daily activity recorded by a well-established triaxial accelerometer.

This will be a single-blinded randomized trial, with subject randomization stratified by age and baseline activity level. Subjects will be randomized to one of three groups: 1) A control group receiving usual care, 2) a group receiving only feedback with associated encouragement about their daily activity, and 3) an intervention group that will receive health coaching with an associated individualized home exercise program.

The study will consist of a 3 month intervention period and a 6 month follow-up/ retention period (total study enrollment period of 9 months). The primary study endpoint is Medtronic device-measured daily activity. All study endpoints will be assessed at baseline, 3 months, and 9 months. The investigators who are conducting study measurements will be blinded to group assignment.

Using a previously established minimum clinically important difference (MCID) of 1.08 hours per day for improvement in daily activity (effect size=1.54) as measured by Medtronic ICDs/CRTs, a total of 8 subjects per group would be needed to achieve a statistical power (1-β) of 0.80 (two-tailed, α=0.05) for a between-groups comparison utilizing two groups. Therefore, depending on the observed effect size in the proposed study, utilizing 3 groups with approximately 10 subjects in each group should provide adequate statistical power for a between-groups comparison with 3 groups.

Statistical analyses will be conducted to meet the planned study objectives. With regard to intervention effects, one way analysis of variance with planned contrasts will be used to examine between-group differences for each of the continuous variables [Patient Activity, Kansas City Cardiomyopathy Questionnaire (KCCQ), Patient Health Questionnaire (PHQ-9), six-minute walk test (6MWT), 30 second timed chair rise (30-s TCR), heart rate variability, Optivol Fluid Index]. If the data do not meet the requisite assumptions, the Kruskal-Wallis analysis of variance by ranks will be used. Baseline to 3 months data will be used to assess immediate intervention effects and to 9 month follow-up will be used to assess retention effects.

With regard to concurrent validity of the Medtronic Patient Activity measurement, the Pearson correlation coefficient will be calculated between the daily Patient Activity (minutes per day) and two Actigraph parameters: daily activity count and steps per day. Correlation coefficients will be calculated for the baseline, 3-month, and 9-month monitoring periods to provide a greater number of sampling days. Correlation coefficients will also be calculated for changes in daily activity measurements between baseline and 3 months and baseline and 9 months to determine concurrent validity of change in daily activity measurements.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of heart failure with subsequent placement of a Medtronic® ICD or Cardiac Resynchronization Therapy (CRT) device at least 6 months prior to study enrollment
* New York Heart Association Functional Class II to III symptoms on optimal medical therapy

Exclusion Criteria:

* Any comorbid medical disease that would prevent safe participation in an individualized exercise program such as severe osteo-, rheumatoid-, and gout-related arthritis, unstable angina, exercise-induced arrhythmias, uncontrollable diabetes, or atrial fibrillation with rapid ventricular rate in the preceding 30 days.
* Recent (<6 weeks) or planned (<6 months) major cardiovascular events or procedures
* Current participation in a regular exercise training program
* HF due to severe, uncorrected primary valvular disease, congenital heart disease, or obstructive cardiomyopathy
* Adults unable to consent (e.g. cognitively impaired), pregnant women, and prisoners

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in Medtronic Implanted Device Patient Activity Measure | Change from baseline to 3 and 9 months

SECONDARY OUTCOMES:
Change in ActiGraph Daily Activity | Change from baseline to 3 and 9 months
Change in Six-Minute Walk Test | Change from baseline to 3 and 9 months
Change in 30 Second Timed Chair Rise | Change from baseline to 3 and 9 months
Change in Kansas City Cardiomyopathy Questionnaire | Change from baseline to 3 and 9 months
Change in 9 Item Patient Health Questionnaire | Change from baseline to 3 and 9 months
Change in Health Care Utilization | Change from baseline to 3 and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Shoemaker, DPT, PhD, Principal Investigator — Grand Valley State University
Locations (1):
- Spectrum Health Heart and Lung Specialized Care Clinic, Grand Rapids, Michigan, United States